CLINICAL TRIAL: NCT03189849
Title: Farms, Animals and Adolescents: Reinforcing the Microbiome
Acronym: FAARM
Status: Completed | Type: Observational
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Other Study IDs: 2017-0154
Record Dates: First submitted 2017-06-01; First posted 2017-06-16 (Actual); Last update posted 2017-10-26 (Actual); Status verified 2017-10

CONDITIONS: Healthy
Keywords: Farming environment

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study will be an observational study of children who attend summer camp at the Heartland Farm Sanctuary (HFS). The investigators are exploring whether time-limited exposure to a traditional farming environment will improve children's overall health and general well-being.

DETAILED DESCRIPTION:
The overarching hypothesis for this study is that urban children exposed on a time-limited basis to a traditional farming environment will show increased beneficial bacteria in the gut microbiome and enhanced emotional well-being. Secondary hypotheses are that 1) increased presence of farm-derived immunoregulatory micro-organisms in the nose (indicating exposure) will be associated with measures of emotional well-being and prosocial behavior. To test these hypotheses, 40 urban children ages 7-13 years will be studied prior to and following a 1, 2, or 3-week camp experience at the Heartland Farm Sanctuary summer camp program in Verona, WI. Assessments for behavior (via questionnaires), gut microbiota composition and function (via stool) and presence in the body of farm-derived immunoregulatory micro-organisms (via nasal swab) will be assessed at baseline (2 weeks before the start of camp and the weekend before camp starts), immediately following the child's 1, 2, or 3-week camp experience and at 1 month following completion of the camp experience. Importantly, this assessment schedule will allow the investigators to assess the longevity of any observed physical or behavioral changes induced by exposure to the farming environment.

ELIGIBILITY:
Inclusion Criteria for Children:

* Males and females ages 7-13 years
* Able to attend camp at Heartland Farm Sanctuary for either 1, 2, or 3 consecutive weeks (if not consecutive, but within a 4-week period, this is allowable)
* In generally good health
* Have not taken antibiotics in the four weeks prior to when their first baseline set of samples will be collected
* Have not attended camp at HFS or regular volunteer activities at HFS in the past year (participation in previous summer HFS camp is permissible)
* Able to understand the nature of the study and able to provide assent
* Able to communicate in English with study personnel.
* Willing to commit to participating in the study and doing the home collection of samples.

Exclusion Criteria for Children:

* Individuals who will not be able to collect the samples for any reason, including planned vacations, unwillingness, or inability. (Note - children who are attending either 2 or 3 weeks of camp and who take a break in between weeks of camp will be allowed to participate if their full two or three-week camp exposure occurs within a 4-week period).
* Plan to attend camp during the fall (i.e. during their month 1 month follow-up)
* Children living in farming environments prior to camp participation
* Children with more than an average of one exposure per week to farm animals, livestock, horses
* Individuals currently on any antibiotic therapy or who will require chronic and/or periodic antibiotic treatment during the study period.
* Subject has a medical condition or disorder that

  * Is unstable, or:
  * Could interfere with the accurate assessment of safety or efficacy of the clinical assessments, including individuals with any:
  * Current participation in any clinical trial that might impact results of this one, which includes participation in another clinical trial where any experimental drugs are being taken as well as studies / drug trials with agents that might affect mood and or the gastrointestinal tract.
* Reasonable likelihood for non-compliance with the protocol for any other reason, in the opinion of the Investigator, prohibits enrollment of subject into the study.

Inclusion Criteria for Parents/Guardians:

* Parent or legal guardian of a child attending HFS summer camp and participating in this study
* Willing to assist the child in the collection of samples as necessary
* Willing to answer questionnaire about their child's participation in the study
* Able to communicate in English with study personnel

Exclusion Criteria for Parents/Guardians:

* Unwilling to assist their child in collection of the samples for this study
* Unwilling to answer questionnaire about their child's participation in the study
* Unable to communicate in English with study personnel

Ages: 7 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: This study will enroll up to 40 children ages 7-13 who attend either 1, 2, or 3 weeks of camp at Heartland Farm Sanctuary. In addition, parents whose children participate in the study will be asked to answer questionnaires about their child.
Sampling Method: Non-Probability Sample
Enrollment: 11 (Actual)
Dates: Start 2017-05-10 (Actual); Primary Completion 2017-09-30 (Actual); Study Completion 2017-09-30 (Actual)

PRIMARY OUTCOMES:
Change in microbiota alpha diversity from baseline to immediately post-camp. | Immediately post-camp
Change in microbiota beta diversity from baseline to immediately post-camp. | Immediately post-camp
Change in the mean scores in the WHO-5 from baseline to immediately post camp. | Immediately post camp
Change in the mean scores in the EmQue-CA from baseline to immediately post camp. | Immediately post camp
Change in the mean scores in the PSC-35 from baseline to immediately post camp. | Immediately post camp
Change in the mean scores in the Youth PSC from baseline to immediately post camp. | Immediately post camp

SECONDARY OUTCOMES:
Change in microbiota alpha diversity from baseline to month 1. | 1 month post-camp
Change in microbiota beta diversity from baseline to month 1. | 1 month post-camp
Change in the mean scores in the WHO-5 from baseline to month 1. | 1 month post-camp
Change in the mean scores in the EmQue-CA from baseline to month 1. | 1 month post-camp
Change in the mean scores in the PSC-35 from baseline to month 1. | 1 month post-camp
Change in the mean scores in the Youth PSC from baseline to month 1. | 1 month post-camp

CONTACTS AND LOCATIONS:
Locations (1):
- University of Wisconsin-Madison, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No